CLINICAL TRIAL: NCT04941092
Title: Clinical Outcomes and Characteristics of Critically Ill Patients With Influenza and COVID-19 Induced ARDS: a Retrospective, Matched Cohort Study
Brief Title: Comparison of ARDS COVID-19 (WHO) vs ARDS Influenza in the ICU
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Lev VOLKOV, Dr, Central Hospital, Nancy, France
Other Study IDs: 2021PI076
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: ARDS; COVID-19 Acute Respiratory Distress Syndrome; Influenza
Keywords: ards
MeSH Terms: conditions — Influenza, Human; Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with ARDS induced by SARS CoV 2
  Interventions: Other: no intervention
- patients with ARDS induced by influenza
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, retrospective comparison

SUMMARY:
Since the beginning of the SARS CoV 2 pandemia, the SARS CoV 2 was frequently compared with the seasonal influenza virus. However, few studies compared patients presenting acute respiratory distress syndrome (ARDS) induced by these viruses, with results being discordant. Our study means to compare mortality and morbidity of patients hospitalized in an intensive care unit (ICU) with ARDS induced by SARS CoV-2 and seasonal influenza.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in ICU
* under mechanical ventilation
* presenting an ARDS according to the Berlin definition
* induced by either influenza or SARS CoV 2

Exclusion Criteria:

* pregnant women
* mechanical ventilation>48 hours before admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized in Intensive Care Unit Hopital Central, Regional University Hospital of Nancy, France
  - hospitalized between 2009 and 2019 if influenza and in 2020 if SARS CoV 2
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
mortality | at 28 days

SECONDARY OUTCOMES:
length of stay in ICU | at 28 days
length of mechanical ventilation | at 28 days
length of vasopressors | at 28 days
length of extrarenal epuration | at 28 days
amount of drugs for sedation | at 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France